CLINICAL TRIAL: NCT02535936
Title: Cortical Plasticity in Spastic Diplegia After Selective Dorsal Rhizotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Manish Narendra Shah, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-15-0335
Record Dates: First submitted 2015-08-25; First posted 2015-08-31 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Spastic Diplegia
Keywords: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3Tesla MRI with DTI-MRI and rsfcMRI (Other): Patients will receive 2 post-operative MRI's with DTI and rsfcMRI at 2 months and 12 months.
  Interventions: Procedure: 3Tesla MRI with DTI-MRI and rsfcMRI under general anesthesia

INTERVENTIONS:
Procedure: 3Tesla MRI with DTI-MRI and rsfcMRI under general anesthesia — 2 post-operative MRI's at 2 months and 12 months

SUMMARY:
The purpose of this study is to characterize the cortical connectivity changes in the brain of spastic diplegic children after Selective Dorsal Rhizotomy.

DETAILED DESCRIPTION:
To establish the structural changes in the corticopyramidal tract using diffusion tractography imaging (DTI) due to selective dorsal rhizotomy and compare the resting state functional connectivity(rsfcMRI) temporal latency differences of spastic diplegics for Selective Dorsal Rhizotomy.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosis with Spastic Diplegia and having Selective Dorsal Rhizotomy surgery

Exclusion Criteria:

* No Selective Dorsal Rhizotomy surgery

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-08; Primary Completion 2030-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Fractional Anisotropy as assessed by brain MRI with diffusion tractography imaging (DTI) sequences | Baseline and 12 months
  This measure will be used to assess changes in the lower extremity fibers corticopyramidal tract after Selective Dorsal Rhizotomy (SDR).
Change in Mean Diffusivity as assessed by brain MRI with diffusion tractography imaging (DTI) sequences | Baseline and 12 months
  This measure will be used to assess changes in the lower extremity fibers corticopyramidal tract Selective Dorsal Rhizotomy (SDR).
Change in Radial Diffusivity as assessed by brain MRI with diffusion tractography imaging (DTI) sequences | Baseline and 12 months
  This measure will be used to assess changes in the lower extremity fibers corticopyramidal tract after Selective Dorsal Rhizotomy (SDR)
Change in Axial Diffusivity as assessed by brain MRI with diffusion tractography imaging (DTI) sequences | Baseline and 12 months
  This measure will be used to assess changes in the lower extremity fibers corticopyramidal tract after Selective Dorsal Rhizotomy (SDR)

CONTACTS AND LOCATIONS:
Overall Officials: Manish N Shah, MD, Principal Investigator — UTHealth Medical School
Locations (1):
- UTHealth & Children's Memorial Hermann Hospital, Houston, Texas, United States